CLINICAL TRIAL: NCT06388863
Title: Evaluation of the Efficacy and Safety of Fecal Microbiota Transplantation for Parkinson's Disease Patients With Constipation
Brief Title: Evaluation of the Efficacy and Safety of Fecal Microbiota Transplantation for Constipation in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B2024-002
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT capsule group (Experimental): Participants will be given 6 FMT capsules twice a week for 24 weeks. The FMT capsules derived from healthy donors.
  Interventions: Drug: Healthy donor-derived FMT capsule
- Placebo capsule group (Placebo Comparator): Participants will be given 6 placebo capsules twice a week for 24 weeks. Placebo capsules are identical in appearance and smell as FMT capsules but contain milk powder.
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: Healthy donor-derived FMT capsule — Participants will be treated with healthy donor-derived fecal microbiota transplantation in the form of oral capsules.
  Arms: FMT capsule group
Drug: Placebo capsule — Capsules whose appearance and smell are identical as FMT capsules but contain milk powder
  Arms: Placebo capsule group

SUMMARY:
Participants will be allocated to FMT group or placebo group at a 1:1 ratio. For interventional group, patients will be given six FMT capsules twice a week for 24 weeks. Placebo capsules are identical in appearance and smell but contain milk powder. At each follow-up visits, participants complete specific scales to assess improvement in constipation, emotion and quality of life. Besides, fecal samples are collected for metagenomics and metabolomics sequencing and blood samples are tested peripheral concentration of levodopa.

DETAILED DESCRIPTION:
This prospective, double-blind, randomised, placebo-controlled study aims to evaluate efficacy and safety of fecal microbiota transplantation for constipation in Parkinson's disease. Participants will be given either FMT capsules or placebo capsules at a ratio of 1:1. For experimental group, patients will be given six FMT capsules twice a week for 24 weeks. Placebo capsules are identical in appearance and smell but contain milk powder. After 24-week treatment, participants complete specific scales to assess improvement in constipation, other PD symptoms, emotion and quality of life. Besides, fecal samples are collected for metagenomics and metabolomics sequencing and blood samples are tested peripheral concentration of levodopa.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who fulfill Chinese diagnostic criteria for PD (2016 edition), aged 40-75 years;
2. PD Hoehn-Yahr stage 1-3
3. Participants who have at least 2 of the following symptoms in the past 3 months and the symptoms have been present for at least 6 months: ① More than 25% of defecations are laborious; ② More than 25% of defecations consist of hard or lumpy stools; ③ More than 25% of defecations are accompanied by a sensation of incomplete evacuation; ④ More than 25% of defecations are accompanied by a sensation of anorectal obstruction; ⑤ More than 25% of defecations require manual assistance; ⑥ Less than 3 spontaneous bowel movements per week.
4. Have taken a stable dose of anti-Parkinson drugs, antidepressants and antipsychotics for at least 1 month;
5. Absence of red flags such as weight loss, hematochezia and exclusion of other diagnosis;
6. Have signed the informed consent and agree to participate in this study;

Exclusion Criteria:

1. Parkinsonism-plus syndrome;
2. Stroke, brain trauma or epilepsy;
3. Have undergone surgery intervention due to PD;
4. Pregnant, planning pregnancy or lactating;
5. Psychiatric disorder or unable to cooperate with treatment and follow-up visit;
6. Immunodeficiency or treatment with immune-modulating medication;
7. Have undergone any abdominal surgery, with the exception of appendectomy, cholecystectomy, caesarean section and hysterectomy;
8. Presence of uncontrolled diabetes, hypertension, thyroid disease or other systemic disease;
9. Use of probiotics or antibiotics within 1 month prior to study entry;
10. Presence of severe diseases related to heart, brain, kidney and lung or concomitant malignancies;

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate of constipation in Parkinson's Disease (PD) | at week 24
  Efficacy index is calculated based on Wexner score. Efficacy index ≥30% is defined as response.

SECONDARY OUTCOMES:
Change from baseline PD symptoms at week 5, week 13 and week 24 | at baseline and week 5, week 13 and week 24
  PD symptoms are assessed via Unified Parkinson's Disease Rating Scale (UPDRS), PD Hoehn-Yahr grade, Non-Motor Symptoms Questionnaire (NMSQ). Change in PD symptoms is obtained by evaluating theses scales at baseline and week 5, week 13 and week 24.
Change from baseline anxiety at week 5, week 13 and week 24 | at baseline and week 5, week 13 and week 24
  Self-rating Anxiety Scale (SAS) is used to evaluate anxiety in PD patients, with a score ranging from 25 to 100. Higher score indicates higher level of anxiety. Change in SAS score is obtained by evaluating the scale at baseline, week 5, week 13 and week 24.
Change from baseline depression at week 5, week 13 and week 24 | at baseline and week 5, week 13 and week 24
  Self-rating Depression Scale (SDS) is used to evaluate depression in PD patients, with a score ranging from 25 to 100. Higher score indicates higher level of depression. Change in SDS score is obtained by evaluating the scale at baseline, week 5, week 13 and week 24.
Change from baseline quality of life at week 5, week 13 and week 24 | at baseline and week 5, week 13 and week 24
  Parkinson's disease Questionnaire (PDQ-39) is used to assess quality of life in PD patients. Higher score indicates worse life quality. Change in PDQ-39 score is obtained by evaluating the scale at baseline, week 5, week 13 and week 24.
Change from baseline drug concentration of levodopa in peripheral blood at week 13 and week 24 | at baseline, week 13 and week 24
  Blood samples are collected and tested for drug concentration of levodopa in peripheral blood
Change from baseline fecal microbiota based on metagenomics sequencing at week 5, week 13 and week 24 | at baseline, week 5, week 13 and week 24
  Fecal samples are collected at baseline, week 5, week 13 and week 24. Change in fecal microbiota is measured by metagenomics.
Change from baseline fecal metabolites based on non-targeted metabolomics at week 5, week 13 and week 24 | at baseline, week 5, week 13 and week 24
  Fecal samples are collected at baseline, week 5, week 13 and week 24. Change in fecal metabolites is measured by non-targeted metabolomics.

CONTACTS AND LOCATIONS:
Overall Officials: Shengdi Wu, Principal Investigator — Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No